CLINICAL TRIAL: NCT00490906
Title: Comparison of Bone Effects With Copaxone and Interferon in Multiple Sclerosis: A Pilot Study
Brief Title: Comparison of Bone Effects With Copaxone and Interferon in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Nancy Hammond, MD (Other)
Collaborators: Kansas City Area Life Sciences Institute, Inc. (Other)
Responsible Party: Sponsor-Investigator, Nancy Hammond, MD, Assistant Professor, Director Comprehensive Epilepsy Center, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: KCALSI-06-01
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Multiple Sclerosis; Low Bone Density
Keywords: MS (Multiple Sclerosis)
MeSH Terms: conditions — Multiple Sclerosis; Bone Diseases, Metabolic | interventions — Glatiramer Acetate; Interferon beta-1a; Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients receive Copaxone
  Interventions: Drug: Copaxone
- 2: Patients receive interferons
  Interventions: Drug: Interferon-beta 1a; Drug: Interferon-beta 1b

INTERVENTIONS:
Drug: Copaxone — 20 mg, subcutaneous injections, taken daily
  Other Names: Glatiramer acetate
  Groups: 1
Drug: Interferon-beta 1a — 30 mcg injected intramuscularly, once weekly
  Other Names: Avonex
  Groups: 2
Drug: Interferon-beta 1b — .25 mg/day, taken every other day, subcutaneous injections
  Other Names: Betaseron
  Groups: 2

SUMMARY:
The purpose of this study is to determine if certain drugs commonly used to treat multiple sclerosis have an effect on bone health.

DETAILED DESCRIPTION:
There will be 60 female patients with MS at University of Kansas Medical Center (KUMC). They will be split into two groups: a Copaxone group and an Interferon (Avonex, Rebif, or Betaseron) group. Each group will be composed of 30 women matched for menopausal status. Each subject will be given a questionnaire assessing risk factors for low bone density. All patients will have a determination of an Expanded Disability Status Scale (EDSS), height and weight, medical history, and fracture history. All patients will undergo hip and spine dual x-ray absorptiometry (DEXA) and will have labs drawn to determine serum 25 hydroxyvitamin D, parathyroid hormone, ionized calcium, estradiol, bone-specific acetyl phosphatase, osteocalcin, and C-peptides.

ELIGIBILITY:
Inclusion Criteria:

* Female, age > 18
* Able to understand and give informed consent
* Relapsing remitting multiple sclerosis (RRMS)
* Treatment with interferons or Copaxone for at least one year prior to study entry

Exclusion Criteria:

* Known osteoporosis
* History of hypercalcemia
* Currently pregnant
* History of primary hyperparathyroidism, hyperthyroidism, or hypothyroidism
* Unstable medical condition
* Ongoing use of bisphosphonates

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants must be female with clinical diagnosis of multiple sclerosis and have been using either Copaxone or interferon injections for the past 1 or more years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Hammond, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - General Clinical Research Center, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas